CLINICAL TRIAL: NCT03682874
Title: Identifying Novel Aging Targets for Treatment of Delirium
Acronym: INNOVATE
Status: Terminated | Type: Observational
Why Stopped: Inability to recruit during COVID-19
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00052417
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-03

CONDITIONS: Delirium; Dementia Alzheimers; Respiratory Failure
MeSH Terms: conditions — Delirium; Alzheimer Disease; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The long-term goal of this research program is to improve understanding of the mechanistic link between Alzheimer's disease (AD) neuropathology, acute delirium, and cognitive impairment following acute respiratory failure. In this pilot study, the study team will establish a prospective cohort of older patients with acute respiratory failure and obtain data on delirium duration, AD imaging and CSF biomarkers, and cognitive outcomes following critical illness.

DETAILED DESCRIPTION:
The study team will recruit patients with no known history of dementia for enrollment into the cohort during their hospital stay for acute respiratory failure. The cohort will undergo testing including cognitive testing, MRI imaging, lumbar puncture for cerebrospinal fluid (CSF) analysis at 3 months following hospital discharge. The study will examine the association of delirium duration during the hospital stay and cognitive impairment at 3 month follow-up with CSF levels of amyloid- β42, tau, and phospho-tau. Measures of delirium will also be related with structural/functional MRI dependent measures. The goal is to design a larger prospective cohort study to evaluate the relationship between AD imaging and CSF biomarkers with delirium and post-ICU cognitive impairment. The results of this pilot study with provide important information with regard to future study design including: (1) ratio of eligible to recruited patients (2) retention rate; (3) safety and feasibility of protocol; and (4) preliminary effect size estimates.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 55 years
* Anticipated ICU stay of at least 48 hours
* Delirium during ICU stay defined as CAM-ICU positive on at least two occasions at least 12 hours apart within 72 hours.

Exclusion Criteria:

* Diagnosis of dementia in electronic medical record at time of ICU admission
* Blindness, deafness, or inability to understand English as this prevents ICU delirium assessment
* Cognitive impairment prior to hospitalization (inability to follow instructions/comply with study/sign consent)
* Score of > 3.30 on Informant Questionnaire of Cognitive -Decline in the Elderly (IQCODE)[34]. Questionnaire will be given to family member or legally authorized representative.
* Pregnancy/lactating/breastfeeding
* Legally incapacitated: Prisoner/Ward of State
* History of prior large vessel cerebrovascular accident (CVA)
* History of neurologic disorder prior to ICU admission including multiple sclerosis, Parkinson disease, epilepsy, amyotrophic lateral sclerosis (ALS), Guillain-Barre Syndrome (GBS)
* Psychiatric illness including schizophrenia, bipolar disorder, depression with psychotic features
* Not expected to survive 24 hours
* Judgment of investigator that subject participation could jeopardize subject health/safety or integrity of study
* Active malignancy requiring treatment in the prior 6 months
* Inability to return for study procedures
* Inability to obtain consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We propose to recruit older patients with acute respiratory failure requiring mechanical ventilation admitted to the medical ICU of an academic medical center, Wake Forest Baptist Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Structural/functional MRI dependent measures | 2-5 months after hospital discharge
  gray matter volume
Structural/functional MRI dependent measures | 2-5 months after hospital discharge
  cerebral blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Palakshappa, MD, Principal Investigator — Wake Forest
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No